CLINICAL TRIAL: NCT07210099
Title: The Effect of Short-term Supplementation of OliPhenolia® on Fat Oxidation in Recreationally Active Volunteers.
Brief Title: The Effect of Short-term Supplementation of OliPhenolia® on Fat Oxidation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Principal Investigator, Justin Roberts, Professor, Anglia Ruskin University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ETH2425-5668
Record Dates: First submitted 2025-06-03; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: FatMax; Fat Oxidation; Polyphenols; Caffeine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 2 main experimental groups in a double-blinded manner. Following completion of the first round of testing, those participants consuming OliPhenolia will return after a 1 week wash out period and repeat the process but taking placebo, and vice versa. Therefore all participants will have consumed either test product or placebo. For the pre-follow up test beverage, participants will be randomly assigned to either placebo or caffeine in block manner. This exploratory study will only involve a single cross over.
Who Masked: Participant, Investigator
Masking Description: Supplements (product, placebo and product and product + caffeine) will be provided in a randomized, double-blinded manner. Both the participants and research testers will be masked from knowing the specifics of the supplement intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OliPhenolia® plus placebo beverage (Experimental): OliPhenolia® is to be consumed twice daily, away from food and separated by ≥4 hours, for a period of 8 days.
  Note each serving of OliPhenolia® is a volume equivalent to ≤1.0mg∙kg-1 of Hydroxytyrosol.
  At the follow up test participants will also be provided with a 150mL placebo (microcrystalline cellulose at a dose of 6mg/kg) beverage pre-exercise.
  Interventions: Dietary Supplement: Concentrated olive fruit water; Dietary Supplement: Placebo beverage
- Placebo product plus placebo beverage (Placebo Comparator): A taste and appearance matched placebo will be used within this research, conforming to the recipe utilised in previously published OliPhenolia® research. Recipe as follows; equal ratio [1:1:1] of prune juice, diet cola, and tonic water. The placebo formula will be provided in matched 28mL sterilised jars provided order to match OliPhenolia® original packaging.
  At the follow up test participants will also be provided with a 150mL placebo (microcrystalline cellulose at a dose of 6mg/kg) beverage pre-exercise.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Placebo beverage
- OliPhenolia® +Caffeine (pre workout) (Experimental): OliPhenolia® is to be consumed twice daily, away from food and separated by ≥4 hours, for a period of 8 days.
  Note each serving of OliPhenolia® is a volume equivalent to ≤1.0mg∙kg-1 of Hydroxytyrosol.
  For the pre workout beverage this will be a single serve drink (150mL) containing flavoured water with 6mg/kg anhydrous caffeine based on previous research. The product will only be used pre-exercise as a single bolus.
  Interventions: Dietary Supplement: Concentrated olive fruit water; Dietary Supplement: Anhydrous caffeine
- Placebo +Caffeine (pre workout) (Active Comparator): A taste and appearance matched placebo will be used within this research, conforming to the recipe utilised in previously published OliPhenolia® research. Recipe as follows; equal ratio [1:1:1] of prune juice, diet cola, and tonic water. The placebo formula will be provided in matched 28mL sterilised jars provided order to match OliPhenolia® original packaging.
  For the pre workout beverage this will be a single serve drink (150mL) containing flavoured water with 6mg/kg anhydrous caffeine based on previous research. The product will only be used pre-exercise as a single bolus.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Anhydrous caffeine

INTERVENTIONS:
Dietary Supplement: Concentrated olive fruit water — Supplementation of OliPhenolia twice daily for eight days. Dose equivalent to ≤1.0mg∙kg-1 of hydroxytyrosol.
  Other Names: OliPhenolia
  Arms: OliPhenolia® +Caffeine (pre workout); OliPhenolia® plus placebo beverage
Dietary Supplement: Placebo — Placebo matched for taste and appearance consumed twice daily for eight days in the equivalent volume to the experimental product.
  Arms: Placebo +Caffeine (pre workout); Placebo product plus placebo beverage
Dietary Supplement: Anhydrous caffeine — A single bolus of flavoured water (150mL) containing 6mg/kg anhydrous caffeine taken as a pre-exercise beverage
  Arms: OliPhenolia® +Caffeine (pre workout); Placebo +Caffeine (pre workout)
Dietary Supplement: Placebo beverage — A single bolus of flavoured water (150mL) containing 6mg/kg microcrystalline cellulose
  Arms: OliPhenolia® plus placebo beverage; Placebo product plus placebo beverage

SUMMARY:
There is current research interest in the use of fruit and plant-based food products containing high levels of natural antioxidants and their impact on exercise, which may be particularly beneficial for recreationally or low-active populations. One such product is an olive extract drink (called OliPhenolia®) produced by Fattoria La Vialla (an organic farm based in Northern Italy) and commercially available for the general public. Whilst previous research from the investigators (at Anglia Ruskin University) using this product has demonstrated potential antioxidant benefits and reduced oxygen cost during aerobic exercise, there are to date no studies investigating whether the short-term consumption of OliPhenolia® can benefit fat oxidation during exercise or whether such effects can be further enhanced employing a pre workout caffeinated beverage.

Therefore the aim of this study is two-fold:

i) to assess the impact of short-term supplementation (8 days) of OliPhenolia® relative to body mass on fat oxidation during aerobic cycling exercise in comparison to placebo in healthy recreationally active volunteers; and ii) whether potential benefits of OliPhenolia® on fat oxidation are enhanced with a pre-workout caffeinated beverage in comparison to placebo in healthy recreationally active volunteers.

DETAILED DESCRIPTION:
This exploratory study will involve initial recruitment of approximately 30-40 healthy volunteers to undertake an initial study briefing pre-screening health questionnaire, informed written consent and familiarisation to exercise equipment, before returning to the human physiology laboratory at Anglia Ruskin University on a separate occasion (Visit 1) to undertake a standard exercise test for maximal fitness capacity.

Following this, Visit 2 will see participants undertake a standard fat oxidation exercise test (aerobic exercise on a cycle ergometer) to ascertain maximal fat oxidation (Fatmax) with increasing exercise intensity, as well as a steady state exercise bout (30mins at FATmax).

After this participants will begin a short-term (8 days) supplementation period of either OliPhenolia or Placebo before returning for a follow up fat oxidation assessment (Visit 3) as above. Fat oxidation will be assessed by standard respiratory measures (breath to breath for oxygen and carbon dioxide). On the follow up test (Visit 3), a pre-exercise workout drink will be provided containing either caffeine flavoured water or placebo. This is to assess whether fat oxidation can be enhanced from short-term polyphenol supplementation (OliPhenolia) with or without additional caffeine prior to exercise.

Participants will therefore be randomised into 1 of 4 groups for this study (Placebo product for 8 days + placebo beverage at follow up; Oliphenolia for 8 days + placebo beverage at follow up; and OliPhenolia for 8 days plus caffeinated beverage at follow up; and placebo product for 8 days plus caffeinated beverage at follow up).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, UK based, above 21 years of age with a body mass index (BMI) >18 and <30 kg·m2 determined during baseline testing

  * Considered to be recreationally active i.e. approximately 150mins of general physical activity/ exercise per week (meeting the WHO physical activity guidelines); and a VO2peak (fitness) score >20 and <50 mL·kg-1·min-1 determined during baseline testing.
  * No known history (including family history) of heart abnormalities, hypertension, coronary heart disease or diabetes (determined from pre-study health screen questionnaire).
  * Not currently suffering from any musculoskeletal injury, or any other reason that may prevent participation in cardiovascular exercise.
  * Have not suffered from recent viral infections ie: influenza (defined within the prior 2 months).
  * Not taking any prescribed or over-the-counter medication which may influence exercise training (with the exception of inhalers for exercise induced asthma or contraceptive pill).
  * Not consuming or prepared to refrain from consumption, any commercial supplementation which conflicts with the study parameters ie: antioxidants.
  * No known allergy or intolerance to olives or prune/grape juice, or any known side effects from caffeine ingestion.

Exclusion Criteria:

* If any of the above criteria is not met.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Maximal fat oxidation (g/min) | Pre and post main intervention (8 days)
  Assessment of total fat oxidation from stochiometrics (based on oxygen and carbon dioxide breath to breath measurements during exercise)

SECONDARY OUTCOMES:
Expired oxygen (L/min) | Pre and post main intervention (8 days)
  Assessment of oxygen cost based on expired air analysis during submaximal exercise

CONTACTS AND LOCATIONS:
Overall Officials: Justin D Roberts, Professor, Principal Investigator — Anglia Ruskin University
Locations (1):
- Cambridge Centre for Sport and Exercise Sciences, Anglia Ruskin University,, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No